CLINICAL TRIAL: NCT03335280
Title: 68Ga-citrate PET/MR Imaging for the Evaluation of Glioma in Adults
Brief Title: 68Ga-citrate PET/MR Imaging for Glioma
Status: Terminated | Type: Observational
Why Stopped: Low Accrual
Sponsor: Susan Chang (Other)
Collaborators: American Brain Tumor Association (Other)
Responsible Party: Sponsor-Investigator, Susan Chang, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: 181016; NCI-2020-00335 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-09-18; First posted 2017-11-07 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive for PTEN deletion: Confirmed by immunohistochemistry of tissue biopsy
  Interventions: Drug: 68Ga-citrate PET/MR
- Negative for PTEN deletion: Confirmed by immunohistochemistry of tissue biopsy
  Interventions: Drug: 68Ga-citrate PET/MR

INTERVENTIONS:
Drug: 68Ga-citrate PET/MR — Study participants will undergo the 68Ga-citrate PET/MR imaging after all screening and baseline assessments have been completed. Patient shall begin imaging between 120 and 360 minutes after the injection of the radiopharmaceutical. Coverage for the scan will extend from the patient's vertex to the neck. The entire imaging study will take roughly 90 minutes.

SUMMARY:
This is a prospective, single center, open-label study in adult patients with presumed World Health Organization (WHO) grade 3 or 4 glioma who will be undergoing surgical resection as standard of care. In some cases, patients will have had biopsy. Study participants will undergo 68Ga-citrate Positron Emission Tomography / magnetic resonance (PET/MR) prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) grade 3 or 4 glioma planning to undergo surgery
* Age >= 18 yrs.
* Karnofsky performance status of >= 60
* Ability to understand a written informed consent document, and the willingness to sign it.

Cohort A:

- Positive for Phosphatase and Tensin Homolog (PTEN) deletion, confirmed by immunohistochemistry of tissue biopsy

Cohort B:

- Negative for PTEN deletion, confirmed by immunohistochemistry of tissue biopsy

Exclusion Criteria:

* Contraindications to Positron Emission Tomography (PET) imaging (e.g. pregnant or breast-feeding woman)
* Contraindications to magnetic resonance (MR) imaging (e.g. pacemakers, metallic implants, etc.)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with WHO grade 3 or 4 glioma planning to undergo surgery with availability of immunohistochemistry of tissue
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-04-24 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Maximum standardized uptake value (SUVmax) | 1 day
  The location and extent of 68Ga-citrate uptake will be compared to both same day magnetic resonance imaging (MRI) and subsequent pathology. SUVmax will be the outcome of interest and summarized with descriptive measures. SUVmax will be compared via a two-sided two-sample equal-variance t-test between those patients positive for PTEN deletion and those negative for PTEN deletion.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03335280/ICF_000.pdf